CLINICAL TRIAL: NCT06517498
Title: Disease Burden and Living Situation of Patients With Facioscapulohumeral Muscular Dystrophy
Status: Recruiting | Type: Observational
Sponsor: Xi'an Jiaotong University (Other)
Collaborators: Chinese Organization for Rare Disorders (Unknown); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Principal Investigator, Wenjing Ji, Associate Professor, Xi'an Jiaotong University
Other Study IDs: XJTU-CDSP_02
Record Dates: First submitted 2024-07-09; First posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Muscular Dystrophy, Facioscapulohumeral
Keywords: Facioscapulohumeral Muscular Dystrophy; Disease Burden; Quality of Life; Living Situation
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients With Facioscapulohumeral Muscular Dystrophy: No intervention will be administered
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention will be conducted

SUMMARY:
The goal of this observational study is to learn the patient journey, disease burden, living situation, quality of life and etc. in patients with Facioscapulohumeral Muscular Dystrophy in all sex/gender and age groups. The main questions it aims to answer are:

1. What's the patient journey of patients with Facioscapulohumeral Muscular Dystrophy?
2. How does Facioscapulohumeral Muscular Dystrophy burden the patients?
3. How's the quality of life of patients with Facioscapulohumeral Muscular Dystrophy?

Patients with Facioscapulohumeral Muscular Dystrophy will be asked to:

1. fill a questionnaire.
2. be interviewed and answer questions about their illness experience, economic burden, quality of life and etc.

Medical experts on Facioscapulohumeral Muscular Dystrophy will be asked to be interviewed and answer questions about understanding on the disease and the patients.

DETAILED DESCRIPTION:
Study Objective This observational study aims to comprehensively understand the patient journey, disease burden, living situation, and quality of life in individuals diagnosed with Facioscapulohumeral Muscular Dystrophy (FSHD). The study encompasses all sex/gender and age groups to provide a holistic view of the disease's impact.

Research Questions

The study focuses on answering the following key questions:

1. What is the patient journey of individuals with Facioscapulohumeral Muscular Dystrophy?
2. How does Facioscapulohumeral Muscular Dystrophy burden the patients?
3. What is the quality of life of patients with Facioscapulohumeral Muscular Dystrophy?

Methodology

To gather comprehensive data, participants will be engaged in two main activities:

1.Questionnaire Completion: Participants will fill out a detailed questionnaire designed to capture quantitative data on their health status, symptoms, treatments received, and the impact of FSHD on their daily lives. The questionnaire will also collect demographic information and other relevant background data.

2.In-Depth Interviews with patients with Facioscapulohumeral Muscular Dystrophy: They will undergo semi-structured interviews conducted by trained researchers. These interviews will delve into the personal experiences of living with FSHD, including:

1. Illness Experience: Participants will describe their journey from initial symptoms to diagnosis and ongoing management of the disease.
2. Economic Burden: Discussions will cover the financial impact of FSHD, including costs related to medical care, treatments, and any income loss due to the inability to work.
3. Quality of Life: Interviews will explore the effects of FSHD on various life domains, such as physical health, mental well-being, social relationships, and overall life satisfaction.

3.In-Depth Interviews with medical experts on Facioscapulohumeral Muscular Dystrophy: They will undergo semi-structured interviews conducted by trained researchers. These interviews will delve into their understanding on the disease and the patients.

Expected Outcomes The study aims to generate a detailed understanding of the multifaceted impact of FSHD on patients' lives. By examining the patient journey, disease burden, and quality of life, the study seeks to identify gaps in current healthcare provisions and areas where additional support may be needed. This information will be valuable for healthcare providers, policymakers, and patient support organizations in improving care and support for individuals with FSHD.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed as Facioscapulohumeral Muscular Dystrophy

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will focus on individuals diagnosed as Facioscapulohumeral Muscular Dystrophy in all sex and age groups.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
EQ-5D | 1 year
  EQ-5D questionnaires will be used to measure the quality of life of the patients. The questionnaires consist of two main parts: Descriptive System and Visual Analog Scale. Descriptive System includes Mobility, Self-Care, Usual Activities, Pain/Discomfort and Anxiety/Depression, each with 5 levels for adults and 3 levels for children. Visual Analog Scalerequires patients to rate their overall health on a scale from 0 to 100, where 0 represents "the worst health you can imagine" and 100 represents "the best health you can imagine." In the end, an index value will be calculated that reflects the patient's overall health status.
Anxiety Level | 1 year
  The Self-Rating Anxiety Scale will be used to measure the anxiety level of the patients. It consists of 20 items, each describing a common symptom of anxiety. Each item is rated on a 4-point Likert scale. The total score ranges from 20 to 80. In doing so, the anxiety level of the patients can be screened.
Economic Burden | 1 year
  Questions will designed to explore the economic burden of the patients. Questions include direct and indirect medical costs over the past year, annual incomes, accumulated treatment costs and debts. Each questions include 7 levels. Besides, whether they have public health insurance and commercial insurance will be asked to discover how much the costs can be covered.
Disease Burden | 1 year
  Questions will designed to explore the disease burden of the patients. Questions include the influence of the disease on respiratory system, dry eyes, whistle, deglutition, speaking and walking. Each question contains 5 levels.

CONTACTS AND LOCATIONS:
Overall Officials: Wenjing Ji, PhD, Principal Investigator — Xi'an Jiaotong University
Locations (1):
- Health Science Center of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared